CLINICAL TRIAL: NCT02022228
Title: Dual Trigger With GnRH Agonist and Human Chorionic Gonadotropin for Final Oocyte Maturation in Patients at High Risk of Ovarian Hyperstimulation Syndrome in GnRH Antagonist Protocol
Brief Title: Dual Trigger to Reduce Ovarian Hyperstimulation Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chenshiling (Other)
Collaborators: National Natural Science Foundation of China (Other Government); Comprehensive Strategic Cooperation Project of Guangdong Province and Chinese Academy of Science (Other); Guangzhou Science and Technology Program key projects (Other); National Key Basic Research Development Plan of China (Unknown)
Responsible Party: Sponsor-Investigator, Chenshiling, Professor, M.D., Ph.D., Nanfang Hospital, Southern Medical University
Organization: Nanfang Hospital, Southern Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Dual Trigger
Record Dates: First submitted 2013-12-15; First posted 2013-12-27 (Estimated); Last update posted 2013-12-27 (Estimated); Status verified 2013-10

CONDITIONS: Infertility and at High Risk of OHSS
Keywords: Ovarian Hyperstimulation Syndrome; Luteinizing Hormone; Polycystic Ovarian Syndrome; Ovarian Yield; Ovarian Maturity; Gonadotropin Releasing Hormone Agonist; Human Chorionic Gonadotropin
MeSH Terms: conditions — Infertility; Ovarian Hyperstimulation Syndrome; Polycystic Ovary Syndrome | interventions — Triptorelin Pamoate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 0.2mg triptorelin and 500 IU hCG (Experimental): Patients were triggered with 0.2mg triptorelin and 500 IU hCG
  Interventions: Drug: triptorelin; Drug: hCG
- 0.2mg triptorelin and 1000 IU hCG (Experimental): Patients were triggered with 0.2mg triptorelin and 1000 IU hCG
  Interventions: Drug: triptorelin; Drug: hCG

INTERVENTIONS:
Drug: triptorelin — 0.2 mg triptorelin, ih
  Other Names: triptorelin: Diphereline
Drug: hCG — 1000 IU hCG, im
  Arms: 0.2mg triptorelin and 1000 IU hCG
Drug: hCG — 500IU hCG, im
  Arms: 0.2mg triptorelin and 500 IU hCG

SUMMARY:
Gonadotropin releasing hormone (GnRH) agonist is sufficient for triggering final oocyte maturation in GnRH antagonist protocol and can significantly reduce incidence of ovarian hyperstimulation syndrome (OHSS) in high-risk patients.

However, lower oocyte yield was reported in patients with lower luteinizing hormone (LH) level post trigger with single injection of GnRH agonist, which might be related to the shorter duration and lower amount of LH induced by GnRH agonist.

Our aim is to study dual trigger with GnRH agonist and human chorionic gonadotropin (hCG) for preventing OHSS and maintaining clinical outcome in high risk patients who receive controlled ovarian stimulation in GnRH antagonist protocol.

ELIGIBILITY:
Inclusion Criteria:

* patients with polycystic ovarian syndrome
* patients with polycystic ovarian morphology on ultrasound
* patients who previously experienced an ovarian stimulation cycle, with a high response to gonadotrophins

Exclusion Criteria:

* patients undergoing coasting
* patients with past ovarian surgery

Max Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 200 (Estimated)
Dates: Start 2012-07; Primary Completion 2015-12 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
clinical pregnancy rate per transfer cycle | 1month post embryo transfer
numbers of patients having OHSS | 2 weeks post trigger with dual GnRHa
oocyte yield | oocyte retrieval day (34 to 38 hours post trigger with GnRHa and hCG)
  Oocyte yield was defined as the ratio of the total number of collected oocytes to the number of follicles measuring ≥10 mm on the day of oocyte retrieval.
Oocyte maturity | 24 hours post oocyte retrieval day
  Oocyte maturity was defined as the ratio of metaphase II (MII) oocytes to the number of collected oocytes in the patients undergoing with intracytoplasmic sperm injection (ICSI).

SECONDARY OUTCOMES:
serum luteinizing hormone level 12 hours post trigger | 12 hours post trigger
serum hCG level 12 hours post trigger | 12 hours post trigger
fertilization rate | 48 hours post IVF/ICSI
  Fertilization rate was defined as the ratio of normal fertilized oocytes (2PNs) to the number of oocytes used for fertilization (i.e. the denominator in IVF in calculating fertilization rate is all oocytes recovered, but in ICSI it is calculated using only the number of MII oocytes).
implantation rate | 1 month post embryo transfer

CONTACTS AND LOCATIONS:
Overall Officials: Shi-Ling Chen, M.D., Ph.D., Study Chair — Nanfang Hospital, Southern Medical University
Locations (1):
- Center for Reproductive Medicine, Department of Gynecology and Obstetrics, Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong, China